CLINICAL TRIAL: NCT02803541
Title: Does a Mainstream Summer Camp Experience Improve Pediatric Kidney Patients' Physical Fitness and Self Concept?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Albert Einstein College of Medicine (Other); YMCA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-1416
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2017-10

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; exercise; pediatrics; summer camp
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 12 day mainstream summer camp experience (Experimental): The 12 day mainstream camp experience involves increased exercise from baseline at home. Can this exercise and peer contact improve physical endurance as measured by the 6 minute walk test and self concept as measured by a modified Harter scale
  Interventions: Behavioral: 12 day mainstream summer camp experience

INTERVENTIONS:
Behavioral: 12 day mainstream summer camp experience — see arm description

SUMMARY:
Purpose: Most children and adolescents with chronic kidney disease (CKD) have much less physical endurance than their age matched peers, are at high risk for premature cardiovascular disease, and have a poor self image in part due to limited peer contact. Sustained exercise in adults with CKD improves endurance and decreases cardiovascular risk. Minimal data exists in pediatric CKD patients. This study will show whether 12 days of increased exercise at a summer camp will improve endurance as measured by the distance walked in 6 minutes and self concept as measured by a short standardized questionaire (Harter scale).

The study will occur at the Frost Valley YMCA in the Catskills where in 2, 12 day sessions a total of 25-30 kidney campers are mainstreamed in the general camp population of about 500.

Mainstreaming means that the kidney camper will live in a cabin with 8-10 age matched peers and participate as much as possible in all camp activities with their bunkmates. The kidney program at Frost Valley provides hemo and peritoneal dialysis, as well as caring for children with less advanced CKD and post transplant.

Participants will have activity measured before and duringcamp by wearing a pedometer. The distance walked in 6 minutes (a 6 minutewalk test) will be measured at onset and completion of the 12 day camp experience. A standardized questionaire on self concept will also be administered at the onset and completion of camp.

DETAILED DESCRIPTION:
BACKGROUND:

Children and adolescents with CKD have high rates of hospitalization, and those with End-Stage Renal Disease (ESRD) have a remaining life expectancy of about 20 years with increased risk of premature death due to cardiovascular disease. Most have much less physical endurance than their age matched peers with the degree of underperformance loosely correlated with the severity of their renal disease. Cardiovascular disease, chronic inflammation, anemia, low muscular strength and/or bone disease are among the factors considered responsible for the poor physical conditioning. However, the investigators hypothesize that the most important cause is inactivity caused by a varying combination of parental 'protection', limited or poor peer inaction, and patient choice. In addition, children who require chronic hemodialysis have an enforced 10-14 hours weekly of enforced inactivity. Cardiovascular morbidity is commonly associated with chronic kidney disease and physical endurance is a measure of cardiovascular health. In addition many children with chronic kidney disease demonstrate poor self-concept, in part related to their lack of physical endurance and limited peer contact.

Multiple studies of adults with chronic kidney disease have documented poor physical conditioning and function. Over the past decade, many studies have demonstrated in adults with CKD a significant benefit of regular exercise on physical fitness, walking capacity, blood pressure, and health related quality of life. Several small studies have shown a modest improvement in children and adolescents with CKD but these studies have had high drop-out rates and problematic compliance.

A 2012 study by Akber et al using pedometer measurements showed that over a 7 day period, children, adolescents, and young adults with CKD (n=44) on average walked about 50% less than expected using data collected by NHANES as a standard. Females walked less than males and older children were less active than younger children. On a 6 minute walk test, males scored < 2 standard deviation below the expected mean and females <4 standard deviation below the mean. There was no measured difference between stage of CKD, dialysis, or transplant status.

In 1975 the Ruth Gottscho Kidney Foundation partnered with the Albert Einstein College of Medicine and the Frost Valley YMCA to develop the first summer camp program capable of performing hemodialysis and caring for children with chronic kidney disease. One of the guiding principles of this program is that kidney campers (as well as some children with other chronic illnesses) are mainstreamed in with the general camp population and participate in the same activities as their age matched peers. Each summer, there are 4 two week camp session with about 500 campers attending each session. The program has run each summer since 1975, and the enrollment of kidney campers has varied from 25 to 50 each summer. The Frost Valley YMCA is located in the Catskill Mountains approximately 120 miles from New York City and is spread over about 2000 acres.

Informal observation of the kidney campers indicates that many show improved physical endurance during their camp stay, and a study done early in the program's history demonstrated an improved self-esteem. , A study using the Piers Harris test of self-concept evaluated 24 chronic dialysis children during the Summer of 1976 and compared them to 76 regular campers. On arrival at camp the dialysis campers had a lower self-concept than the regular campers (P<.01). The same children were evaluated at the end of camp. Both groups improved their self-concept (P<0.02) but the dialysis campers showed greater improvement. (P<0.01) This study was presented at the 1977 Clinical Dialysis and Transplant Forum.

The investigators hypothesize that during their time at camp the kidney campers will improve their physical endurance and their self-concept; which will be assessed objectively through physical fitness/function and psychometric assessments. The investigators hope to do this in a way that interferes as little as possible with the camp experience yet is educational and fun for the kidney campers and their peers.

The ultimate objective of this pilot study is to increase awareness that children with CKD should be physically active, can enjoy being part of a program with their peers, and may benefit physically and mentally from it.

METHODS:

This pilot study designed in close collaboration between the UNC Kidney Center and the UNC Department of Exercise Science and will occur during the first two 12 day camp sessions at the Frost Valley YMCA during the Summer of 2016.

Campers range in age from 8 to 17 years. Each kidney camper and age matched healthy controls (bunkmates) will be provided with a pedometer before camp arrival and will be asked to wear it throughout each day in the week before camp in order to record their physical activity level. Participants will also be asked to record screen time during the week prior to beginning the camp. Participants will be asked to wear the pedometer during their camp stay, except during waterfront activities, and the data recorded. The investigators hope to enroll all kidney campers (estimate 25-40 individuals) and approximately 70-100 control campers.

The Omron 321 pedometer was chosen because it retains seven-days of data, is inexpensive, and has been previously shown to be a valid and reliable indicator of physical activity.

On the day of, or the first day after camp arrival, each kidney camper along with his/her bunkmates will be asked to complete a 6 minute walk test (6MWT). A standardized chart to self-report their perceived exertion at the end of the walk will be used. Pulse upon completion of the 6MWT and 1 minute later will be measured. Each child will wear a portable pulse oximeter during the walk. The investigators hypothesize that the kidney campers will increase their activity at camp compared to their activity at home as measured by the pedometer, and also that they will be able to ambulate further as measured by the 6MWT with less perceived exertion and possibly lower post 6MWT pulse rate at the end of the camp session as compared to the beginning of camp.

The 6MWT test was chosen as the primary test measurement in consultation with the Exercise Science Department faculty and camp administrative staff as there is considerable normative data in healthy children, it is non-invasive, and its administration can easily fit into the camp program.

Having the kidney campers participate with their bunkmates in the 6MWT will provide motivation for campers to perform at as high a level as possible, yet not single the kidney campers out as special or specifically as research subjects. Research data will be collected only for those campers for whom consent/assent has been obtained.

Similarly, data for the control campers will be instructive as to whether a relatively short period of increased activity (12 days) will allow measured changes in their 6MWT.

In order to be time efficient and fit in with the camp environment, rather than the standard 6MWT which is classically done in a hallway between 2 cones separated by 20 meters, the campers will walk (not run) along the camp circle from approximately the laundry area to Biscuit Hall (modified 6MWT). This is a relatively level paved path (net elevation rise ~15 feet) about 1500 feet in distance and is estimated to take the average camper about 6 minutes. Any who reach Biscuit Hall earlier, will do laps around Biscuit until the 6 minutes is up. The course will be carefully measured and marked so that distances achieved will be accurately ascertained.

The 6MWT will be repeated in the identical fashion shortly before the end of the camp session, at approximately the same time of day.

Any child who becomes unusually fatigued during the modified 6MWT, will be encouraged to rest until he or she is ready to continue.

A short standardized survey to measure self-concept will be given to the kidney campers and to control campers to be completed upon arrival and shortly prior to leaving camp using the Harter Self Perception Profile for Children (SPPC).

Camp physical forms will be used to determine age, weight, and height for control campers and be directly measured for the kidney campers.

STATISTICS The primary data collected will be the distance traveled on the 6MWT. Each child will serve as his/her own control for paired t-test analysis. Secondary data, which will emphasize the kidney campers, will be perceived exertion and self concept. In both groups, if possible, correlations will be drawn between activity levels prior to camp, performance on the 6MWT, and measurement of self-concept. Also, group analyses will be done with comparisons to previously published standard data.

As this is a pilot project and little data exists on the activity levels of children with kidney disease and no similar study has ever been done, it is difficult to predict what changes in activity will be seen. Consequently power calculations are not provided. Similarly, most studies of exercise use periods considerably longer than 12 days, so it is possible that 12 days is insufficient to see a measureable change in the 6MWT.

Although all campers in the bunk or village will be asked to participate in the 6MWT, only data from those campers whose families have provided consent and campers who have provided assent will be used for analysis. If sufficient non-kidney campers participate, data can be analyzed in a similar manner to measure the impact of the camp experience on their physical fitness and self-concept. In this situation, data regarding screen time pre camp as well as the pedometer measurements pre-camp may be instructive.

ELIGIBILITY:
Inclusion Criteria:

* All kidney campers attending the Frost Valley YMCA and age matched otherwise healthy campers who provide consent

Exclusion Criteria:

* none

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk distance | Baseline , Day 12
  The change in 6MWT distance measured in feet from Baseline to Day 12

SECONDARY OUTCOMES:
Change in SPPC scores from Baseline to Day 12 | Baseline, Day 12
  Harter Self Perception Profile for Children (SPPC) consists of 36 items representing five domains of self-esteem (i.e., scholastic competence, social acceptance, athletic competence, physical appearance, and behavioral conduct, as well as global self-worth). Each SPPC item consists of two opposite descriptions. Respondents choose the best fitting description indicating whether the description is "somewhat true" or "very true" for them. Items are scored on a four-point scale with a higher score reflecting a more positive view of oneself. The scale will be modified since the scholastic competence domain will not be included because the study is occurring during summer school vacation.
Exertion perception from the 6 minute walk | Baseline, day 12
  The Exertion Perception will be self-evaluated using the BORG scale at the end of the 6 minute walk. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort
Is 12 days of increased exercise long enough to see changes in endurance? | Baseline, day 12
  Will there be improvement in the 6 MWT from baseline to day 12 in the kidney campers. A similar analysis will be done for the nonkidney campers if sufficient number of campers are recruited

CONTACTS AND LOCATIONS:
Overall Officials: William Primack, MD, Principal Investigator — Nephrology
Locations (1):
- Frost Valley YMCA, Claryville, New York, United States

IPD SHARING:
Plan to Share IPD: No